CLINICAL TRIAL: NCT01183442
Title: Effects of Vitamin D Supplementation in Coronary Artery Disease Patients With Postchallenge Hyperglycemia and Vitamin D Deficiency on Endothelial Function and Insulin Sensitivity
Brief Title: Vitamin D Supplementation in CAD and Postchallenge Hyperglycemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: unable to recruit
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENM-DA012
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease; Postprandial Hyperglycemia; Vitamin D Deficiency
Keywords: endothelial function; insulin sensitivity
MeSH Terms: conditions — Coronary Artery Disease; Hyperglycemia; Vitamin D Deficiency; Insulin Resistance | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D (Oleovit®) (Active Comparator): vitamin D drops
  Interventions: Drug: vitamin D
- Placebo (Placebo Comparator): placebo drops
  Interventions: Drug: vitamin D

INTERVENTIONS:
Drug: vitamin D — orally administered 2800 IU of vitamin D or placebo daily
  Other Names: vitamin d (Oleovit®)

SUMMARY:
The main aim of the investigation is to clarify, whether vitamin D supplementation in coronary artery disease patients with vitamin D deficiency and postchallenge hyperglycemia has an impact on endothelial dysfunction and parameters of insulin sensitivity and beta-cell function.

DETAILED DESCRIPTION:
An improvement of endothelial dysfunction as a cardiovascular surrogate parameter could be translated in a reduced risk for future cardiovascular events, which is of major interest, since patients with postchallenge hyperglycemia face a significantly higher cardiovascular risk than patients with normal glucose tolerance. Furthermore an improvement in insulin sensitivity and/or beta-cell function would identify vitamin D as an important strategy for the prevention of type 2 diabetes. In consideration of the rapidly increasing prevalence of diabetes and the failure of current prevention strategies this could be an important, safe and cheap way to support ongoing lifestyle modifying programs. Our study of course investigates surrogate cardiovascular and insulin sensitivity parameters. Assuming a beneficial effect of vitamin D in our study, this concept would have to be proven in further large outcome as well as diabetes prevention trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75
* Postchallenge hyperglycemia (2h-whole blood glucose value in oral glucose tolerance test above 119 mg/dl, normal fasting glucose)
* Angiographically verified coronary artery disease (>50% stenosis)
* Serum 25-OH- vitamin D < 20 ng/ml in winter/spring/autumn and <25 ng/ml during june-september
* Stable antihypertensive therapy in the last 3 month

Exclusion Criteria:

* Acute coronary syndrome or cerebrovascular event within the previous 1 month
* BMI > 40 kg/m²
* Serum creatinine >2.5 times the upper limit of normal
* GOT or GPT > 3 times the upper limit of normal
* Heart failure > NYHA class II
* Uncontrolled hypertension (>160/100 mmHg)
* New onset of statins, ACE-inhibitors or ARBs within the previous 4 weeks
* History of urolithiasis
* Hypercalcaemia
* Major psychiatric disorders
* Ongoing treatment with spironolactone, canrenoate, eplerenone, amiloride, triamterene and aliskiren.
* Treatment with antipsychotic drugs
* Regular significant antioxidants, vitamins or protein supplementation
* Immunosuppressive therapy
* Glucocorticoid therapy
* Ongoing chemotherapy
* Pregnancy
* Any other disease with an estimated life expectancy below 1 year.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
endothelial dysfunction | 1 year
  Changes in endothelial dysfunction (peripheral artery tone (PAT) and biochemical)

SECONDARY OUTCOMES:
insulin resistance and beta-cell function | 1 year
  Changes in indices for insulin resistance and beta-cell function

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University of Graz, Graz, Austria
Locations (1):
- Dept. of Internal Medicine, Medical University of Graz, Graz, Austria